CLINICAL TRIAL: NCT01055743
Title: A Randomized, Controlled Trial of Fluorouracil Implants Regional Chemotherapy During the Surgical Treatment for Early Stage Hepatocellular Carcinoma
Brief Title: The Effect of Fluorouracil Implants Regional Chemotherapy During the Surgical Treatment for Early Stage Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Shuqun Cheng, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009PHC001
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Early Stage Hepatocellular Carcinoma
Keywords: Fluorouracil Implants; Hepatocellular carcinoma; Radical resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radical resection + Fluorouracil Implants (Experimental)
  Interventions: Procedure: Radical resection; Drug: Fluorouracil Implants
- Radical resection (Active Comparator)
  Interventions: Procedure: Radical resection

INTERVENTIONS:
Procedure: Radical resection — Radical resection of hepatocellular carcinoma
Drug: Fluorouracil Implants — Implanted during the surgical treatment
  Arms: Radical resection + Fluorouracil Implants

SUMMARY:
This study will assess the clinical efficacy and safety of fluorouracil implants regional chemotherapy during the surgical treatment for early-stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of stage I hepatocellular carcinoma
* Child-Pugh class A, B
* Radical resection is feasible
* Patients with adequate renal, hepatic, and hematologic function
* Written informed consent

Exclusion Criteria:

* Allergic to chemotherapy drugs
* No measurable lesion
* Receive chemotherapy, radiotherapy or biotherapy within 30 days prior to enrollment
* Evidence of serious infection
* Renal or hepatic dysfunction, significant cardiovascular disease
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical benefit of fluorouracil implants regional chemotherapy during the radical resection in early stage hepatocellular carcinoma patients. The primary endpoint is disease-free survival (DFS). | 1, 2, and 3 years

SECONDARY OUTCOMES:
Quality of Life | from baseline to the last visit
Incidence Rate of Complications | 1, 2, and 3 years
Adverse Events | from the beginning of treatment to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Shuqun Cheng, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China